CLINICAL TRIAL: NCT05623319
Title: Phase 2 Trial of Translational Approach to First Line cHemoimmunotherapy Followed by Maintenance With pembrOlizumab and Olaparib in Extensive-Stage Small-Cell Lung CanceR.
Brief Title: Pembrolizumab and Olaparib Treatment of Extensive Small Cell Lung Cancer (ES-SCLC)
Acronym: THOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST162.14
Record Dates: First submitted 2022-10-31; First posted 2022-11-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: SCLC,Extensive Stage
Keywords: SCLC,Extensive Stage; Translational; Liquid Biopsy; Pembrolizumab; Olaparib
MeSH Terms: interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab/Olaparib (Experimental): Patients will be treated with pembrolizumab plus chemotherapy during the Induction Phase. In case of responsive or stable disease, patients will enter the Maintenance Phase and will be treated with pembrolizumab plus olaparib until progression or up to a maximum of 35 cycles.
  Interventions: Drug: Pembrolizumab/Olaparib

INTERVENTIONS:
Drug: Pembrolizumab/Olaparib — Patients will receive pembrolizumab 200 mg 1q21 and chemotherapy -platinum compound (cisplatin 75 mg/m2 or carboplatin area under the curve of 5 mg per milliliter per minute) 1q21 plus etoposide 100 mg/m2 1-3q21- for 4 cycles (Induction Phase). In case of responsive or stable disease, patients will receive pembrolizumab 200 mg 1q21 plus olaparib 300 mg twice daily until progression (Maintenance Phase) or up to a maximum of 35 cycles.

SUMMARY:
This is an open-label, single arm, phase 2 trial enrolling patients with untreated Extensive-Stage Small-Cell Lung Cancer (ES SCLC), with a strong translational attitude.

DETAILED DESCRIPTION:
SCLC is a very aggressive disease with an overall survival (OS) of 12 months in the extensive stage (ES). Platinum-based as the first line of treatment has an overall response rate (ORR) of approximately 70% with a progression-free survival (PFS) of 5.5 months and an OS of almost 10 months. Prophylactic cranial irradiation, performed in order to prevent progression in brain, one of the major sites of recurrence, was associated with an increase in median disease-free survival of 12.0-14.7 weeks and in median OS of 5.4-6.7 months with a 1-year survival rate of 27.1%. At recurrence few therapeutic options are available. In order to improve clinical results, several strategies are under evaluation. Given the strong activity shown in several settings, immunotherapy is studied both as a single agent and in combinations.

Pembrolizumab has shown as maintenance after chemotherapy a PFS of 6.9 months in Programmed Cell Death 1 Ligand 1 (PD-L1) positive patients and as a monotherapy in 2nd and further lines an ORR of 19.3%, with major responses in PD-L1 positive patients and 61% of responders lasting ≥18 months. Recently the addition to standard chemotherapy of atezolizumab in patients with untreated ES-SCLC has led to an improvement of 2 months in OS (12.3 in the combo arms vs. 10.3 months in the control arm) and a slight improvement in PFS (5.2 vs. 4.3 months, respectively), without new safety data. Similarly addition of durvalumab to standard chemotherapy has led to a 2.7 months OS improvement (13 in the combo arms vs. 10.3 months in the control arm) with a relevant improvement in ORR (79.5 vs 70.3% respectively), without any improvement in PFS. Finally pembrolizumab combined with chemotherapy has shown significant improvement in PFS (hazard ratio (HR), 0.75; 95% confidence interval (CI), 0.61-0.91) but not in OS. Finally, considering the role of DNA damage repair systems in the tumorigenesis of SCLC, Olaparib has been also evaluated together with durvalumab in pre-treated ES-SCLC obtaining a clinical benefit of 21.1% and confirmed responses or stable disease for ≥8 months. Tumor responses were observed in all instances in which pretreatment tumors showed an inflamed phenotype. Despite biologic knowledge is growing, no clinically relevant molecular features have been identified. Recent publications in fact have proposed a new classification of SCLC in 3 major subgroups according to the expression of the neuronal basic helix-loop-helix transcription factors achaete-scute homologue 1 (ASCL1), involved in the neuroendocrine characterization, and the neurogenic differentiation factor 1 (NEUROD1). The so-called "classic type" shows expression of ASCL1, the "variant type" expresses NEUROD1 and the third type is negative for both the two previous biomarkers. In terms of gene profiling these subgroups are distinct but without a clear prognostic and predictive role. No driver mutations have been found. Many pathways are under evaluations. In particular Poly(ADP-Ribose) Polymerase (PARP) protein levels are up - regulated in SCLC relative to other lung cancers. In particular, Poly(ADP-Ribose) Polymerase 1 (PARP1) has been found to be highly expressed at both the messenger RNA (mRNA) and protein levels in SCLC samples. Given these data the combination proposed (Induction Phase with platinum/etoposide/pembrolizumab followed by a Maintenance Phase with pembrolizumab/olaparib) may be a new therapeutic option to be explored for patients. Moreover the evaluation of molecular features performed before, during and after this treatment may produce new evidence for further clinical trials.

The primary objective of the study is to evaluate the efficacy of chemo-immunotherapy induction followed by maintenance with pembrolizumab and olaparib in terms of Progression-free Survival (PFS).

Patients with extensive stage (ES) SCLC will receive pembrolizumab 200 mg 1q21 with platinum compound (cisplatin 75 mg/m2 or carboplatin area under the curve of 5 mg per milliliter per minute) 1q21 plus etoposide 100 mg/m2 1-3q21 for 4 cycles (Induction Phase). In case of responsive or stable disease, patients will receive pembrolizumab 200 mg 1q21 plus olaparib 300 mg twice daily until progression (Maintenance Phase) or up to a maximum of 35 cycles.

Patients will be accrued for a period of 24 months and follow-up will continue for a period of 12 months after the last patient is enrolled.

The Kaplan-Meier approach will be used to estimate PFS.

ELIGIBILITY:
The Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Male/female participants who are at least 18 years of age on the day of signing informed consent.
3. Cytologically/histologically confirmed diagnosis of SCLC per the Veterans Administration Lung Study Group (VALG) staging system will be enrolled in this study. Patients must have extensive stage (ES) SCLC defined as Stage IV (T any, N any, M 1a/b/c) by the American Joint Committee on Cancer, Eighth Edition.
4. Possibility of obtaining tissue sample, via a biopsy of the primary tumour or metastatic tumour tissue, within the 6 weeks prior to study entry. An archival biopsy is acceptable as long as there has been no intervening anticancer treatment since the time the biopsy was obtained to enrolment in this clinical study and as long as it was within 6 weeks of study entry. Tissue sample would consist of formalin-fixed, paraffin-embedded tumour tissue blocks, or, from formalin-fixed paraffin-embedded tumor tissue block, at least five re-cut, unstained sections of 5 μM thickness for immunohistochemical analysis and five unstained sections of 10 μM thickness for NGS, presented on slides or cell-block.
5. No prior systemic treatment for ES-SCLC. Patients who have received prior chemo-radiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment free interval of at least 6 months since the last chemotherapy, radiotherapy, or chemoradiotherapy cycle from diagnosis of ES-SCLC.
6. Patients with thoracic radiotherapy clinically indicated (e.g. mediastinal syndrome) could be enrolled providing they receive radiotherapy not before 15 days since the start of the experimental treatment. Patients who received radiation therapy to the lung fields that is > 30 Gy within 6 months of the first dose of trial treatment, will be excluded.
7. Presence of target lesions by RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of registration .
9. Patients with paraneoplastic syndromes can be enrolled if an autoimmune origin can be excluded. Autoimmune origin will be defined according to local practice.
10. Life expectancy ≥12 weeks.
11. Capacity to swallow.
12. Ability to comply with the study protocol, in the investigator's judgment.
13. Have adequate organ function. Specimens must be collected within 10 days prior to the registration day.
14. Negative human immunodeficiency virus (HIV) test at screening.
15. Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
16. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
17. Male participants: Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception.
18. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix F, or
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix F during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
2. Active or history of autoimmune disease or immune deficiency which has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs), including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     * Rash must cover less than 10% of body surface area;
     * Disease is well controlled at baseline and requires only low-potency topical corticosteroids;
     * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months;
     * Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
3. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
4. Prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT interval by Fredericia (QTcF) prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome. In case of significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident), acute events must happen not before than 3 months prior to initiation of study treatment.
7. Major surgical procedure within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.
8. History of malignancy other than SCLC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as, adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, Stage I uterine cancer or non-muscle-invasive urothelial carcinoma (Ta - Tis - T1).
9. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
10. Active infection requiring systemic therapy.
11. Known history of active Bacillus Tuberculosis (TB).
12. Treatment with investigational therapy within 28 days prior to initiation of study treatment.
13. Patient who has received prior therapy with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, anti-Cytotoxic T-Lymphocyte Associated Protein 4 (CTLA-4), anti-OX40, anti-Cluster of Differentiation 137 (CD137), anti-CD27).
14. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2 (IL-2)) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment.
15. Any previous treatment with a PARP inhibitor, including Olaparib.
16. Concomitant use of known strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
17. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
18. Has severe hypersensitivity (≥Grade 3) to pembrolizumab, olaparib and/or any of their excipients.
19. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
20. Known allergy or hypersensitivity to carboplatin or etoposide.
21. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
24. Has had an allogenic tissue/solid organ transplant.
25. A WOCBP who has a positive urine pregnancy test within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 44 months
  Time from registration to the first documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by local site or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 36 months
  Percentage of patients who have a confirmed complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1) during the induction and the maintenance phases of treatment.
Immune-related Objective response rate (irORR). | 36 months
  Percentage of patients achieving a complete response (CR) or partial response (PR), according to immune-modified RECIST 1.1 criteria, during the induction and the maintenance phases of treatment.
Progression free survival (PFS) at 6, 12, and 24 months | About at 6-12-24 months
  Percentage of patients alive and progression-free at 6, 12, and 24 months.
Overall Survival (OS) | 44 months
  Time from registration to death due to any cause
Number of participants experiencing Adverse Events (AEs). | 44 months
  Number of participants discontinuing study drugs due to AEs. Toxicity rate: percentage of patients experiencing a specific adverse event of grade 3-5, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the induction and the maintenance phases of treatment.
PD-L1 analysis | 44 months
  Evaluation of Programmed Cell Death 1 Ligand (PD-L1) expression on biopsy and blood samples collected before, during and after the treatment. It will be investigated the association of this marker with study drugs response, including efficacy and/or adverse events.
DNA damage repair analysis | 44 months
  Evaluation of DNA damage repair (DDR) alterations on biopsy and blood samples collected before, during and after the treatment. It will be investigated the association of this marker with study drugs response, including efficacy and/or adverse events.
Tumor Mutational Burden analysis | 44 months
  Evaluation of Tumor Mutational Burden (TMB) on biopsy and blood samples collected before, during and after the treatment. It will be investigated the association of this marker with study drugs response, including efficacy and/or adverse events.
MicroSatellite Instability analysis | 44 months
  Evaluation of MicroSatellite Instability (MSI) on biopsy and blood samples collected before, during and after the treatment. It will be investigated the association of this marker with study drugs response, including efficacy and/or adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Delmonte, Study Chair — IRCCS IRST
Locations (12):
- Italy (12):
  - UO Oncologia Medica, IRST IRCCS, Meldola, Forlì Cesena
  - Ospedale San Gerardo - ASST Monza, Monza, Monza E Brianza
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Pesaro Urbino
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - UO Oncologia, IRCCS Ospedale Sant'Orsola, AUSL Bologna, Bologna
  - IRCCS Istituto Nazionale Tumori Fondazione "G. Pascale", Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda USL della Romagna - Osp. Santa Maria delle Croci, Ravenna
  - A.O. Arcispedale S. Maria Nuova IRCCS di Reggio Emilia, Reggio Emilia
  - Azienda USL della Romagna - Osp. "Infermi" di Rimini, Rimini
  - Istituti Fisioterapici Ospitalieri - IFO -Ospedale Regina Elena, Roma
  - ASST dei Sette Laghi - Osp. di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: No